CLINICAL TRIAL: NCT06674031
Title: Investigation of Knowledge of Cardiovascular Risk Factors and Perception of Benefits and Barriers to Exercise in Patients with Chronic Kidney Disease
Brief Title: Knowledge of Cardiovascular Risk Factors in Chronic Kidney Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: SBA 23/275
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease(CKD); Renal Transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic kidney disease
- Healthy individuals

SUMMARY:
The aim of this study is to assess knowledge of cardiovascular risk factors, physical activity levels, health literacy and perceptions of benefits and barriers to exercise in patients with chronic kidney disease and compare them with healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease
* Being aged 18-65
* Voluntary participation in the study

Exclusion Criteria:

* Having cognitive problems
* Being illiterate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients and healthy individuals will be included in the study.
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Knowledge of cardiovascular risk factors | 10 minutes
  It will be evaluated Cardiovascular Diseases Risk Factors Knowledge Level scale. The maximum score that can be obtained from the 28-question scale is 28. Higher scores indicate better knowledge of cardiovascular disease.
Exercise benefits/barriers | 10 minutes
  This will be evaluated using exercise benefits/barriers scale. Possible scores on the benefits scale ranged from 29 to 116 points. Higher scores indicate greater benefits.The range of possible scores on the barriers scale was 14 to 54 points. Higher scores indicate fewer perceived barriers.
Physical activity | 5 minutes
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short form. This questionnaire lists activities and asks for estimates of the duration and frequency of each activity in the past week. The durations are multiplied by the MET value for each activity and the results for all items are summed to give an overall physical activity score.

SECONDARY OUTCOMES:
Health literacy | 5 minutes
  It will be evaluated with the Health Literacy Scale-Short Form. The score ranges from 0 to 50, with higher scores indicating better health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)